CLINICAL TRIAL: NCT02710526
Title: A Phase II, Open-label, Partially Randomized, 3 Treatment Groups, Multi-Site Study Assessing Pharmacokinetics After Administration of the Once-Weekly and Once-Monthly, Long-Acting Subcutaneous Injectable Depot of Buprenorphine (CAM2038) at Different Injection Sites in Opioid-Dependent Subjects With Chronic Pain
Brief Title: Phase II Pharmacokinetics Study of CAM2038
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Braeburn Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-15-549
Record Dates: First submitted 2016-03-09; First posted 2016-03-16 (Estimated); Results first posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Opioid Use Disorder; Chronic Pain
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 32 mg CAM2038 weekly (Experimental): Group 1, 32 mg of CAM2038 subcutaneous weekly injection at multiple injection sites
  Interventions: Drug: CAM2038
- 128 mg CAM2038 monthly injection (Experimental): Group 2: 128 mg of CAM2038 subcutaneous monthly injection in the buttocks
  Interventions: Drug: CAM2038
- 160 mg CAM2038 monthly injection (Experimental): Group 3: 24mg sublingual BPN for the first 7 days, and then 160 mg of CAM2038 subcutaneous monthly injection in the buttocks starting on Day 8.
  Interventions: Drug: CAM2038

INTERVENTIONS:
Drug: CAM2038 — Long-Acting Subcutaneous Injectable Depot of Buprenorphine
  Other Names: Buprenorphine

SUMMARY:
Phase II, open label, partially randomized, three treatment group study designed to evaluate the steady state pharmacokinetics of buprenorphine and norbuprenorphine following repeated subcutaneous administrations of CAM2038.

DETAILED DESCRIPTION:
This is a phase II, open label, partially randomized, three treatment group study designed to evaluate the steady state pharmacokinetics of buprenorphine and norbuprenorphine following repeated subcutaneous administrations of CAM2038 weekly and monthly at different injection sites and to evaluate the steady state pharmacokinetics of buprenorphine and norbuprenorphine after repeated subcutaneous administration of CAM2038 monthly in opioid dependent subjects with a history of chronic non cancer pain. The study will involve three phases: Screening, Treatment, and Follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent prior to the conduct of any study related procedures.
2. Male or non pregnant, non lactating female subject, aged 19 to 65 years, inclusive.
3. Body mass index between 19 and 35 kg/m2, inclusive.
4. Current diagnosis of moderate to severe opioid use disorder (according to the DSM 5) or past medical history of opioid use disorder currently being treated with SL BPN.
5. Subject must be taking SL BPN (Subutex® equivalent) 24 mg (Group 1 and Group 2) or ≥24 mg (Group 3) daily for at least 30 days prior to Screening.
6. Subject has a history of moderate to severe chronic non cancer pain.
7. Male and female subjects of childbearing potential must be willing to use a reliable method of contraception during the entire study (Screening visit to Follow-up phone call).
8. Subject must be willing and able to comply with all study procedures and requirements.

Exclusion Criteria:

1. Individuals meeting DSM-V substance use disorder criteria for alcohol, benzodiazepines, central nervous system (CNS) stimulants, or other drugs of abuse (excluding caffeine, tobacco or THC/marijuana).
2. Any clinically significant abnormality on the basis of medical history, vital signs, physical examination, 12-lead electrocardiogram (ECG; Fridericia's corrected QT interval [QTcF] ≥450 msec. for males or ≥470 msec. for females), and laboratory evaluations (including hematology, clinical chemistry, urinalysis at Screening), in the opinion of the Investigator.
3. Significant symptoms, medical conditions, or other circumstances which, in the opinion of the Investigator, would preclude compliance with the protocol, adequate cooperation in the study or obtaining informed consent, or may prevent the subject from safely participating in study, including subjects who are at a risk for gastrointestinal obstruction or paralytic ileus or who have severe respiratory insufficiency, respiratory depression, airway obstruction, gastrointestinal motility disorders, biliary tract disease, severe hepatic insufficiency, planned surgery and prior treatment with monoamine oxidase inhibitors.
4. Use (therapeutic or non-therapeutic) of opioids other than SL BPN.
5. Aspartate aminotransferase (AST) levels > 3 X the upper limit of normal, alanine aminotransferase (ALT), levels > 3 X the upper limit of normal, total bilirubin > 1.5 X the upper limit of normal, or creatinine > 1.5 X upper limit of normal on the Screening laboratory assessments, or other clinically significant laboratory abnormalities, which in the opinion of the Investigator may prevent the subject from safely participating in study.
6. Pregnant or lactating or planning to become pregnant during the study.
7. Diagnosis of, or currently under investigation for, fibromyalgia, complex regional pain syndrome, neurogenic claudication due to spinal stenosis, spinal cord compression, acute nerve root compression, severe or progressive lower extremity weakness or numbness.
8. History of chemotherapy or confirmed malignancy (except basal cell or squamous carcinoma of the skin) within the past 2 years.
9. Clinically significant history of, or current evidence for, suicidal ideation or those who are actively suicidal, as based on the Columbia-Suicide Severity Rating Scale (C-SSRS; grade 4 or 5).
10. Clinically significant history of major depressive disorder that is poorly controlled with medication.
11. Hypersensitivity or allergy to BPN or other opioids, or excipients of CAM2038.
12. Exposure to any investigational drug within the 4 weeks prior to Screening.
13. Participants with a clinically significant history of risk factors of Torsades de Pointes and any existing ventricular tachyarrhythmias such as bigeminy, trigeminy, heart failure, hypokalemia, family history of Long QT Syndrome.
14. On medications that have the potential for prolonging the QT interval or who may require such medications during the course of the study along with clinically significant abnormalities on screening electrocardiogram (ECG) readings as deemed by the investigator.
15. Requires current use of agents that are strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) such as some azole antifungals (e.g., ketoconazole), macrolide antibiotics (e.g., clarithromycin), or protease inhibitors (e.g., ritonavir, indinavir, and saquinavir).
16. Intolerance to venipuncture and/or difficulty with venous access, as per the judgment of the Investigator/research staff.
17. Is an employee of the Investigator or the study site, with direct involvement in the proposed study or other studies under the direction of the Investigator or study site, or is a family member of an employee or of the Investigator.
18. Any pending legal action that could prohibit participation or compliance in the study.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-02; Primary Completion 2017-05-17 (Actual); Study Completion 2017-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Sullivan, Principal Investigator — Parkway Medical Center
Locations (3):
- United States (3):
  - Parkway Medical, Birmingham, Alabama
  - Hassman Research Institute, Berlin, New Jersey
  - The Rivus Wellness & Research Institute, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bjornsson M, Acharya C, Strandgarden K, Tiberg F. Population Pharmacokinetic Analysis Supports Initiation Treatment and Bridging from Sublingual Buprenorphine to Subcutaneous Administration of a Buprenorphine Depot (CAM2038) in the Treatment of Opioid Use Disorder. Clin Pharmacokinet. 2023 Oct;62(10):1427-1443. doi: 10.1007/s40262-023-01288-6. Epub 2023 Aug 16. PMID 37584841

RESULTS

PARTICIPANT FLOW:
Groups:
- 32 mg CAM2038 Weekly: Group 1, 32 mg of CAM2038 subcutaneous weekly injections at multiple injection sites
  CAM2038: Long-Acting Subcutaneous Injectable Depot of Buprenorphine
- 128 mg CAM2038 Monthly Injection: Group 2: 128 mg of CAM2038 subcutaneous monthly injections during Treatment Phase and 32 mg of CAM2038 subcutaneous weekly injections during Safety Extension in the buttocks
  CAM2038: Long-Acting Subcutaneous Injectable Depot of Buprenorphine
- 160 mg CAM2038 Monthly Injection: Group 3: 24 mg SL BPN for the first 7 days and then 160 mg of CAM2038 subcutaneous monthly injections in the buttocks starting on Day 8
  CAM2038: Long-Acting Subcutaneous Injectable Depot of Buprenorphine
Period: Treatment Phase
Arm/Group | 32 mg CAM2038 Weekly | 128 mg CAM2038 Monthly Injection | 160 mg CAM2038 Monthly Injection
Started | 28 | 20 | 18
Completed | 22 | 16 | 12
Not Completed | 6 | 4 | 6
Period: Safety Extension
Arm/Group | 32 mg CAM2038 Weekly | 128 mg CAM2038 Monthly Injection | 160 mg CAM2038 Monthly Injection
Started | 15 | 12 | 0
Completed | 14 | 12 | 0
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 160 mg CAM2038 Monthly Injection: Group 3: 24 mg SL BPN for the first 7 days and then 160 mg of CAM2038 subcutaneous monthly injection in the buttocks starting on Day 8
  CAM2038: Long-Acting Subcutaneous Injectable Depot of Buprenorphine
- Total: Total of all reporting groups
Arm/Group | 32 mg CAM2038 Weekly | 128 mg CAM2038 Monthly Injection | 160 mg CAM2038 Monthly Injection | Total
Number analyzed (Participants) | 28 | 20 | 17 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (10.83) | 48.0 (11.49) | 44.1 (12.23) | 45.3 (11.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 4 | 9 | 27
  Male | 14 | 16 | 8 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 27 | 20 | 17 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 4
  White | 27 | 20 | 13 | 60
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.0 (3.95) | 27.0 (4.25) | 28.3 (3.72) | 26.9 (4.04)

OUTCOME MEASURES:

1. Primary Outcome: AUCss(Area Under the Plasma Concentration-time Curve During a 7-day Dosing Interval at Steady State) for Each Injection Site, i.e., Buttock (Reference), Abdomen, Thigh and Back of Upper Arm for the Evaluable Pharmacokinetic (PKEVAL) Population
Description: AUCss (area under the plasma concentration-time curve during a 7-day dosing interval at steady state) for each injection site, i.e., buttock (reference), abdomen, thigh and back of upper arm-Buprenorphine for the Evaluable Pharmacokinetic (PKEVAL) Population
Time Frame: PK samples were collected at pre-dose and at 0.5, 1, 2, 4, 6, 10, 24, 30, 48, 72, 96, 120 and 168 hours post-CAM2038 q1w for Doses/Weeks 4, 5, 6, and 7.
Population: Evaluable Pharmacokinetic (PKEVAL) Population consisted of all subjects who had sufficient PK data for all 4 randomized injection sites to derive PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- 32 mg CAM2038 Weekly-Buttock: Group 1, 32 mg of CAM2038 subcutaneous weekly injection at Buttock
  CAM2038: Long-Acting Subcutaneous Injectable Depot of Buprenorphine
- 32 mg CAM2038 Weekly-Abdomen: Group 1, 32 mg of CAM2038 subcutaneous weekly injection at Abdomen
  CAM2038: Long-Acting Subcutaneous Injectable Depot of Buprenorphine
- 32 mg CAM2038 Weekly-Thigh: Group 1, 32 mg of CAM2038 subcutaneous weekly injection at Thigh
  CAM2038: Long-Acting Subcutaneous Injectable Depot of Buprenorphine
- 32 mg CAM2038 Weekly-Upper Arm: Group 1, 32 mg of CAM2038 subcutaneous weekly injection at Upper Arm
  CAM2038: Long-Acting Subcutaneous Injectable Depot of Buprenorphine
Arm/Group | 32 mg CAM2038 Weekly-Buttock | 32 mg CAM2038 Weekly-Abdomen | 32 mg CAM2038 Weekly-Thigh | 32 mg CAM2038 Weekly-Upper Arm
Number analyzed (Participants) | 21 | 21 | 21 | 20
ng*h/mL | 700 (27.1) | 657 (27.2) | 613 (36.8) | 591 (33.7)

2. Primary Outcome: Css,av(Average Plasma Concentration During a Dosing Interval at Steady State) for Each Injection Site for the Evaluable Pharmacokinetic (PKEVAL) Population
Description: Css,av (average plasma concentration during a dosing interval at steady state) for each injection site-Buprenorphine for the Evaluable Pharmacokinetic (PKEVAL) Population
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 32 mg CAM2038 Weekly-Buttock | 32 mg CAM2038 Weekly-Abdomen | 32 mg CAM2038 Weekly-Thigh | 32 mg CAM2038 Weekly-Upper Arm
Number analyzed (Participants) | 21 | 21 | 21 | 20
ng/mL | 4.17 (27.1) | 3.91 (27.2) | 3.65 (36.8) | 3.52 (33.7)

3. Primary Outcome: Css,Max (Maximum Observed Plasma Concentration During a Dosing Interval at Steady State) for Each Injection Site.
Description: Css,max (maximum observed plasma concentration during a dosing interval at steady state) for each injection site-Buprenorphine
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 32 mg CAM2038 Weekly-Buttock | 32 mg CAM2038 Weekly-Abdomen | 32 mg CAM2038 Weekly-Thigh | 32 mg CAM2038 Weekly-Upper Arm
Number analyzed (Participants) | 21 | 21 | 21 | 21
ng/mL | 6.87 (37.2) | 6.56 (29.9) | 5.37 (43.6) | 5.69 (43.1)

4. Primary Outcome: Tss,Max (Time to Maximum Concentration at Steady State) for Each Injection Site
Description: Tss,max (time to maximum concentration at steady state) for each injection site-buprenorphine
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | 32 mg CAM2038 Weekly-Buttock | 32 mg CAM2038 Weekly-Abdomen | 32 mg CAM2038 Weekly-Thigh | 32 mg CAM2038 Weekly-Upper Arm
Number analyzed (Participants) | 21 | 21 | 21 | 21
h | 24.0 [0.0 to 72.0] | 24.0 [0.0 to 168] | 24.0 [10.0 to 120] | 24.0 [4.0 to 48.0]

5. Primary Outcome: Area Under the Curve at Steady State (AUC During a 28-day Dosing Interval at Steady State)-Buprenorphine
Description: Area Under the Curve at steady state (AUC during a 28-day dosing interval at steady state)-Buprenorphine for Pharmacokinetic Population
Time Frame: PK samples were collected at pre-dose, 0.5, 1, 2, 4, 6, and 10 hours and at approximately 24, 48, 72,96, 120, 168 (7 days), 240 (10 days), 336 (14 days), 504 (21 days) and 672 (28 days) hours after CAM2038 q4w Dose 4
Population: Pharmacokinetic (PK) Population consisted of all subjects in the Safety population who provided PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- 160 mg CAM2038 Monthly Injection: Group 3: 160 mg of CAM2038 subcutaneous monthly injection in the buttocks
  CAM2038: Long-Acting Subcutaneous Injectable Depot of Buprenorphine
Arm/Group | 128 mg CAM2038 Monthly Injection | 160 mg CAM2038 Monthly Injection
Number analyzed (Participants) | 16 | 12
ng*h/mL | 2610 (41.7) | 3540 (26.1)

6. Primary Outcome: Average Steady State Concentration-Buprenorphine
Description: Average steady state concentration-Buprenorphine-Pharmacokinetic Population
Time Frame: as for outcome 5
Population: Pharmacokinetic (PK) Population consisted of all subjects in the Safety population who provided PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 128 mg CAM2038 Monthly Injection | 160 mg CAM2038 Monthly Injection
Number analyzed (Participants) | 16 | 11
ng/mL | 3.89 (41.7) | 5.27 (26.1)

7. Primary Outcome: Maximum Steady State Concentration-Buprenorphine
Description: Maximum steady state concentration-BuprenorphinePharmacokinetic (PK) Population
Time Frame: as for outcome 5
Population: Pharmacokinetic (PK) Population consisted of all subjects in the Safety population who provided PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 24 mg SL BPN: Group 3: 24 mg SL BPN-daily
Arm/Group | 128 mg CAM2038 Monthly Injection | 160 mg CAM2038 Monthly Injection | 24 mg SL BPN
Number analyzed (Participants) | 16 | 12 | 16
ng/mL | 11.1 (54.1) | 15.4 (52.0) | 11.1 (61.4)

8. Primary Outcome: Time to Maximum Concentration at Steady State-Buprenorphine
Description: Time to maximum concentration at steady state-Buprenorphine Pharmacokinetic (PK) Population
Time Frame: as for outcome 5
Population: Pharmacokinetic (PK) Population consisted of all subjects in the Safety population who provided PK data.
Measure: Median (Full Range); unit: h
Arm/Group | 128 mg CAM2038 Monthly Injection | 160 mg CAM2038 Monthly Injection | 24 mg SL BPN
Number analyzed (Participants) | 16 | 12 | 16
h | 10.0 [1.0 to 48.0] | 24.0 [6.1 to 48.3] | 1.69 [0.00 to 4.07]

9. Primary Outcome: Norbuprenorphine/Buprenorphine Ratios at Maximum Concentration at Steady State
Description: Norbuprenorphine/buprenorphine ratios at maximum concentration at steady state Evaluable Pharmacokinetic (PKEVAL) Population
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | 32 mg CAM2038 Weekly-Buttock | 32 mg CAM2038 Weekly-Abdomen | 32 mg CAM2038 Weekly-Thigh | 32 mg CAM2038 Weekly-Upper Arm
Number analyzed (Participants) | 21 | 21 | 21 | 21
ratio | 0.305 (59.1) | 0.307 (53.9) | 0.366 (60.3) | 0.366 (55.2)

10. Primary Outcome: AUCss(Area Under the Plasma Concentration-time Curve During a 7-day Dosing Interval at Steady State) for Each Injection Site, i.e., Buttock (Reference), Abdomen, Thigh and Back of Upper Arm.
Description: AUCss (area under the plasma concentration-time curve during a 7-day dosing interval at steady state) for each injection site, i.e., buttock (reference), abdomen, thigh and back of upper arm-Norbuprenorphine Evaluable Pharmacokinetic (PKEVAL) Population
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 32 mg CAM2038 Weekly-Buttock | 32 mg CAM2038 Weekly-Abdomen | 32 mg CAM2038 Weekly-Thigh | 32 mg CAM2038 Weekly-Upper Arm
Number analyzed (Participants) | 18 | 17 | 17 | 17
ng*h/mL | 204 (70.5) | 192 (69.0) | 208 (90.9) | 197 (70.1)

11. Primary Outcome: Css,av(Average Plasma Concentration During a Dosing Interval at Steady State) for Each Injection Site
Description: Css,av (average plasma concentration during a dosing interval at steady state) for each injection site-Norbuprenorphine-Evaluable Pharmacokinetic (PKEVAL) Population
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 32 mg CAM2038 Weekly-Buttock | 32 mg CAM2038 Weekly-Abdomen | 32 mg CAM2038 Weekly-Thigh | 32 mg CAM2038 Weekly-Upper Arm
Number analyzed (Participants) | 18 | 17 | 17 | 17
ng/mL | 1.22 (64.3) | 1.15 (69.0) | 1.24 (90.9) | 1.17 (70.1)

12. Primary Outcome: Css,Max (Maximum Observed Plasma Concentration During a Dosing Interval at Steady State) for Each Injection Site.
Description: Css,max (maximum observed plasma concentration during a dosing interval at steady state) for each injection site-Norbuprenorphine-Evaluable Pharmacokinetic (PKEVAL) Population
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 32 mg CAM2038 Weekly-Buttock | 32 mg CAM2038 Weekly-Abdomen | 32 mg CAM2038 Weekly-Thigh | 32 mg CAM2038 Weekly-Upper Arm
Number analyzed (Participants) | 21 | 21 | 21 | 21
ng/mL | 1.85 (74.5) | 1.78 (67.2) | 1.74 (86.7) | 1.84 (78.2)

13. Primary Outcome: Tss,Max (Time to Maximum Concentration at Steady State) for Each Injection Site
Description: Tss,max (time to maximum concentration at steady state) for each injection site-Norbuprenorphine-Evaluable Pharmacokinetic (PKEVAL) Population
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | 32 mg CAM2038 Weekly-Buttock | 32 mg CAM2038 Weekly-Abdomen | 32 mg CAM2038 Weekly-Thigh | 32 mg CAM2038 Weekly-Upper Arm
Number analyzed (Participants) | 21 | 21 | 21 | 21
h | 72.0 [0.0 to 120] | 72.0 [0.0 to 168] | 72.0 [0.5 to 168] | 30.0 [0.0 to 168]

14. Primary Outcome: Norbuprenorphine/Buprenorphine Ratios for Area Under the Curve at Steady State
Description: Norbuprenorphine/buprenorphine ratios for Area Under the Curve at steady state Evaluable Pharmacokinetic (PKEVAL) Population
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | 32 mg CAM2038 Weekly-Buttock | 32 mg CAM2038 Weekly-Abdomen | 32 mg CAM2038 Weekly-Thigh | 32 mg CAM2038 Weekly-Upper Arm
Number analyzed (Participants) | 21 | 21 | 21 | 20
ratio | 0.354 (57.4) | 0.341 (52.5) | 0.355 (54.4) | 0.370 (50.7)

15. Primary Outcome: Area Under the Curve at Steady State (AUC During a 28-day Dosing Interval at Steady State)-Norepinephrine
Description: Area Under the Curve at steady state (AUC during a 28-day dosing interval at steady state)-Norepinephrine-Pharmacokinetic (PK) Population
Time Frame: as for outcome 5
Population: Pharmacokinetic (PK) Population consisted of all subjects in the Safety population who provided PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 128 mg CAM2038 Monthly Injection | 160 mg CAM2038 Monthly Injection
Number analyzed (Participants) | 16 | 11
ng*h/mL | 795 (130.5) | 1590 (55.1)

16. Primary Outcome: Average Steady State Concentration-Norbuprenorphine
Description: Average steady state concentration-Norbuprenorphine-Pharmacokinetic (PK) Population
Time Frame: as for outcome 5
Population: Pharmacokinetic (PK) Population consisted of all subjects in the Safety population who provided PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 128 mg CAM2038 Monthly Injection | 160 mg CAM2038 Monthly Injection
Number analyzed (Participants) | 16 | 11
ng/mL | 1.18 (130.5) | 2.37 (55.1)

17. Primary Outcome: Maximum Steady State Concentration-Norbuprenorphine
Description: Maximum steady state concentration-Norbuprenorphine-Pharmacokinetic (PK) Population
Time Frame: PK samples at pre-dose, 0.5, 1, 2, 4, 6,10 hrs and approx. 24, 48, 72, 96, 120, 168, 240, 336, 504 and 672 hrs after CAM2038 q4w Dose 4 and pre-dose (within 45 mins), 10, 20, 30 and 40 mins, and 1, 1.5, 2, 3, 4, 6, 10, and 24 hrs after SL BPN dose 7
Population: Pharmacokinetic (PK) Population consisted of all subjects in the Safety population who provided PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 24 mg SL BPN: Group 3: 24 mg SL BPN daily
Arm/Group | 128 mg CAM2038 Monthly Injection | 160 mg CAM2038 Monthly Injection | 24 mg SL BPN
Number analyzed (Participants) | 16 | 12 | 16
ng/mL | 2.14 (122.8) | 4.61 (54.5) | 7.92 (75.6)

18. Primary Outcome: Time to Maximum Concentration at Steady State-Norbuprenorphine
Description: Time to maximum concentration at steady state-Norbuprenorphine-Pharmacokinetic (PK) Population
Time Frame: as for outcome 17
Population: Pharmacokinetic (PK) Population consisted of all subjects in the Safety population who provided PK data.
Measure: Median (Full Range); unit: h
Groups:
- 24 mg SL BPN: Group 3: 24mg SL BPN daily
Arm/Group | 128 mg CAM2038 Monthly Injection | 160 mg CAM2038 Monthly Injection | 24 mg SL BPN
Number analyzed (Participants) | 16 | 12 | 16
h | 84.1 [0.50 to 244] | 121 [2.17 to 671] | 1.78 [0.68 to 6.47]

19. Secondary Outcome: Number of Participants With Adverse Events for Both Weekly and Monthly CAM2038
Description: Number of Participants with Adverse Events for Both weekly and monthly CAM2038-Safety Population
Time Frame: 99 days for Group 1, 162 days for Group 2, 127 days for Group 3
Population: Safety Population: included all subjects who received CAM2038
Measure: Number; unit: participants
Arm/Group | 32 mg CAM2038 Weekly | 128 mg CAM2038 Monthly Injection | 160 mg CAM2038 Monthly Injection
Number analyzed (Participants) | 28 | 20 | 17
participants
  Subjects with TEAEs | 14 | 10 | 9
  Subjects with Serious TEAEs | 0 | 0 | 0
  Subjects with suspected to be drug-related TEAEs | 4 | 3 | 2
  Subjects with AEs that resulted in death | 0 | 0 | 0
  Subjects with at least 1 AE | 14 | 10 | 9
  Subjects with mild grade AEs | 3 | 4 | 4
  Subjects with moderate grade AEs | 11 | 5 | 5
  Subjects with severe grade AEs | 0 | 1 | 0
  Subjects with at least 1 injection site TEAE | 3 | 1 | 0
  Subjects with mild grade injection site AEs | 0 | 0 | 0
  Subjects with moderate grade injection site AEs | 3 | 1 | 0
  Subjects with severe grade injection site AEs | 0 | 0 | 0
  Subjects with at least 1 non-injection site AE | 13 | 10 | 9
  Subject with mild grade non-injection site AEs | 3 | 4 | 4
  Subject with moderate grade non-injection site AEs | 10 | 5 | 5
  Subjects with severe grade non-injection site AEs | 0 | 1 | 0
  Subjects with TEAEs that led to drug withdrawn | 0 | 0 | 0

20. Other Pre Specified Outcome: Summary of Average Daily Pain by Week (ITT Population)
Description: Summary of Average Daily Pain, using an 11-point Numerical Rating Scale (NRS) for pain, following repeated subcutaneous administration of CAM2038 weekly and CAM2038 monthly in adult opioid-dependent subjects. 11 point scale ranging from 0-10, with 0 being the least amount of pain to 10 being the worst pain imaginable. (ITT Population)
Time Frame: 99 days for Group 1, 162 days for Group 2, 127 days for Group 3
Population: ITT Population-consisted of all subjects who received at least 1 injection of CAM2038 and provided some efficacy measures. Participants did not always enter pain scores in electronic diaries. Also, participants early terminated during the study and stopped entering scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 32 mg CAM2038 Weekly | 128 mg CAM2038 Monthly Injection | 160 mg CAM2038 Monthly Injection
Number analyzed (Participants) | 28 | 20 | 17
score on a scale
  Baseline: number analyzed (Participants) | 6 | 4 | 16
  Baseline | 5.7 (1.06) | 6.7 (2.28) | 5.0 (2.18)
  Week 1: number analyzed (Participants) | 27 | 19 | 17
  Week 1 | 4.4 (2.37) | 3.4 (2.25) | 4.5 (2.12)
  Week 2: number analyzed (Participants) | 25 | 18 | 15
  Week 2 | 4.0 (2.19) | 3.7 (2.44) | 4.1 (1.52)
  Week 3: number analyzed (Participants) | 24 | 18 | 16
  Week 3 | 3.9 (2.18) | 4.0 (2.59) | 4.5 (1.79)
  Week 4: number analyzed (Participants) | 23 | 18 | 16
  Week 4 | 3.2 (2.08) | 3.9 (2.71) | 4.4 (2.10)
  Week 5: number analyzed (Participants) | 23 | 16 | 15
  Week 5 | 3.3 (2.00) | 3.0 (1.99) | 4.0 (1.84)
  Week 6: number analyzed (Participants) | 22 | 17 | 16
  Week 6 | 3.2 (1.88) | 3.2 (2.39) | 3.7 (1.76)
  Week 7: number analyzed (Participants) | 23 | 17 | 15
  Week 7 | 3.0 (2.01) | 3.7 (2.20) | 4.3 (1.88)
  Week 8: number analyzed (Participants) | 15 | 17 | 14
  Week 8 | 3.5 (1.47) | 3.9 (2.00) | 4.8 (2.04)
  Week 9: number analyzed (Participants) | 14 | 16 | 13
  Week 9 | 3.7 (1.88) | 3.5 (2.27) | 3.7 (2.05)
  Week 10: number analyzed (Participants) | 12 | 15 | 12
  Week 10 | 3.3 (1.50) | 3.3 (1.94) | 4.1 (2.11)
  Week 11: number analyzed (Participants) | 11 | 15 | 11
  Week 11 | 3.9 (1.66) | 3.0 (2.10) | 4.1 (2.23)
  Week 12: number analyzed (Participants) | 10 | 15 | 11
  Week 12 | 3.6 (1.51) | 3.6 (1.98) | 4.4 (2.23)
  Week 13: number analyzed (Participants) | 10 | 15 | 11
  Week 13 | 3.9 (1.63) | 2.8 (2.23) | 3.1 (1.81)
  Week 14: number analyzed (Participants) | 3 | 14 | 10
  Week 14 | 6.0 (3.42) | 3.2 (1.98) | 3.8 (1.80)
  Week 15: number analyzed (Participants) | 0 | 14 | 10
  Week 15 |  | 3.2 (2.16) | 4.1 (1.91)
  Week 16: number analyzed (Participants) | 0 | 12 | 10
  Week 16 |  | 3.9 (2.30) | 4.5 (2.15)
  Week 17: number analyzed (Participants) | 0 | 10 | 3
  Week 17 |  | 4.1 (1.92) | 4.3 (1.44)
  Week 18: number analyzed (Participants) | 0 | 10 | 0
  Week 18 |  | 3.9 (2.46) |
  Week 19: number analyzed (Participants) | 0 | 11 | 0
  Week 19 |  | 4.2 (2.22) |
  Week 20: number analyzed (Participants) | 0 | 9 | 0
  Week 20 |  | 4.4 (1.93) |
  Week 21: number analyzed (Participants) | 0 | 10 | 0
  Week 21 |  | 4.3 (2.06) |
  Week 22: number analyzed (Participants) | 0 | 10 | 0
  Week 22 |  | 4.2 (2.40) |
  Week 23: number analyzed (Participants) | 0 | 1 | 0
  Week 23 |  | 6.0 (NA) — Only one participant entered a score, so no SD. |

21. Other Pre Specified Outcome: Number of Participants With Confirmed Opiate Independence as Confirmed by Negative Urine Toxicology Tests
Description: Number of Participants with confirmed Opiate Independence as confirmed by Negative Urine Toxicology Tests-ITT Population
Time Frame: 99 days for Group 1, 162 days for Group 2, 127 days for Group 3
Population: ITT Population: included all subjects who received at least one dose of CAM2038 and provided some efficacy measures-Note that some patients dropped from the study so the numbers at the baseline may be different from later visits.
Measure: Count of Participants; unit: Participants
Arm/Group | 32 mg CAM2038 Weekly | 128 mg CAM2038 Monthly Injection | 160 mg CAM2038 Monthly Injection
Number analyzed (Participants) | 28 | 20 | 17
Participants
  Baseline | 16 | 12 | 14
  Day 1: number analyzed (Participants) | 25 | 17 | 17
  Day 1 | 13 | 11 | 13
  Day 2: number analyzed (Participants) | 27 | 20 | 17
  Day 2 | 14 | 12 | 15
  Day 3: number analyzed (Participants) | 0 | 0 | 17
  Day 3 |  |  | 15
  Day 4: number analyzed (Participants) | 0 | 0 | 15
  Day 4 |  |  | 13
  Day 5: number analyzed (Participants) | 0 | 0 | 15
  Day 5 |  |  | 13
  Day 6: number analyzed (Participants) | 0 | 0 | 17
  Day 6 |  |  | 15
  Day 7: number analyzed (Participants) | 0 | 0 | 17
  Day 7 |  |  | 15
  Day 8: number analyzed (Participants) | 25 | 17 | 14
  Day 8 | 13 | 12 | 11
  Day 9: number analyzed (Participants) | 0 | 0 | 17
  Day 9 |  |  | 14
  Day 15: number analyzed (Participants) | 25 | 18 | 17
  Day 15 | 11 | 10 | 12
  Day 22: number analyzed (Participants) | 24 | 18 | 17
  Day 22 | 12 | 9 | 9
  Day 23: number analyzed (Participants) | 24 | 0 | 0
  Day 23 | 14 |  |
  Day 24: number analyzed (Participants) | 23 | 0 | 0
  Day 24 | 14 |  |
  Day 25: number analyzed (Participants) | 24 | 0 | 0
  Day 25 | 13 |  |
  Day 26: number analyzed (Participants) | 23 | 0 | 0
  Day 26 | 13 |  |
  Day 27: number analyzed (Participants) | 24 | 0 | 0
  Day 27 | 15 |  |
  Day 29: number analyzed (Participants) | 24 | 17 | 17
  Day 29 | 12 | 9 | 10
  Day 30: number analyzed (Participants) | 24 | 0 | 0
  Day 30 | 9 |  |
  Day 31: number analyzed (Participants) | 24 | 16 | 0
  Day 31 | 11 | 8 |
  Day 32: number analyzed (Participants) | 23 | 0 | 0
  Day 32 | 12 |  |
  Day 33: number analyzed (Participants) | 24 | 0 | 0
  Day 33 | 10 |  |
  Day 34: number analyzed (Participants) | 23 | 0 | 0
  Day 34 | 10 |  |
  Day 36: number analyzed (Participants) | 23 | 17 | 16
  Day 36 | 11 | 9 | 13
  Day 37: number analyzed (Participants) | 23 | 0 | 0
  Day 37 | 10 |  |
  Day 38: number analyzed (Participants) | 21 | 0 | 15
  Day 38 | 11 |  | 11
  Day 39: number analyzed (Participants) | 23 | 0 | 0
  Day 39 | 10 |  |
  Day 40: number analyzed (Participants) | 23 | 0 | 0
  Day 40 | 10 |  |
  Day 41: number analyzed (Participants) | 23 | 0 | 0
  Day 41 | 9 |  |
  Day 43: number analyzed (Participants) | 23 | 16 | 17
  Day 43 | 10 | 10 | 14
  Day 44: number analyzed (Participants) | 23 | 0 | 0
  Day 44 | 9 |  |
  Day 45: number analyzed (Participants) | 22 | 0 | 0
  Day 45 | 9 |  |
  Day 46: number analyzed (Participants) | 23 | 0 | 0
  Day 46 | 9 |  |
  Day 47: number analyzed (Participants) | 22 | 0 | 0
  Day 47 | 9 |  |
  Day 48: number analyzed (Participants) | 22 | 0 | 0
  Day 48 | 9 |  |
  Day 50: number analyzed (Participants) | 25 | 17 | 17
  Day 50 | 8 | 8 | 8
  Day 57: number analyzed (Participants) | 0 | 16 | 17
  Day 57 |  | 10 | 13
  Day 59: number analyzed (Participants) | 0 | 13 | 0
  Day 59 |  | 9 |
  Day 64: number analyzed (Participants) | 0 | 15 | 16
  Day 64 |  | 10 | 12
  Day 66: number analyzed (Participants) | 0 | 0 | 15
  Day 66 |  |  | 12
  Day 71: number analyzed (Participants) | 14 | 16 | 15
  Day 71 | 7 | 9 | 10
  Day 78: number analyzed (Participants) | 0 | 16 | 15
  Day 78 |  | 9 | 12
  Day 85: number analyzed (Participants) | 0 | 16 | 15
  Day 85 |  | 10 | 13
  Day 86: number analyzed (Participants) | 0 | 16 | 0
  Day 86 |  | 9 |
  Day 87: number analyzed (Participants) | 0 | 16 | 0
  Day 87 |  | 9 |
  Day 88: number analyzed (Participants) | 0 | 16 | 0
  Day 88 |  | 9 |
  Day 89: number analyzed (Participants) | 0 | 15 | 0
  Day 89 |  | 9 |
  Day 90: number analyzed (Participants) | 0 | 15 | 0
  Day 90 |  | 8 |
  Day 92: number analyzed (Participants) | 12 | 16 | 12
  Day 92 | 6 | 9 | 9
  Day 93: number analyzed (Participants) | 0 | 0 | 12
  Day 93 |  |  | 9
  Day 94: number analyzed (Participants) | 0 | 0 | 12
  Day 94 |  |  | 9
  Day 95: number analyzed (Participants) | 0 | 14 | 12
  Day 95 |  | 8 | 9
  Day 96: number analyzed (Participants) | 0 | 0 | 12
  Day 96 |  |  | 9
  Day 97: number analyzed (Participants) | 0 | 0 | 12
  Day 97 |  |  | 10
  Day 99: number analyzed (Participants) | 0 | 16 | 11
  Day 99 |  | 10 | 9
  Day 102: number analyzed (Participants) | 0 | 0 | 10
  Day 102 |  |  | 7
  Day 106: number analyzed (Participants) | 0 | 15 | 12
  Day 106 |  | 8 | 9
  Day 113: number analyzed (Participants) | 0 | 18 | 12
  Day 113 |  | 11 | 8
  Day 120: number analyzed (Participants) | 0 | 0 | 17
  Day 120 |  |  | 12
  Day 134: number analyzed (Participants) | 0 | 12 | 0
  Day 134 |  | 5 |
  Day 155: number analyzed (Participants) | 0 | 12 | 0
  Day 155 |  | 7 |

22. Other Pre Specified Outcome: Subject-rated Worst Daily Pain
Description: Subject-rated worst daily pain, using an 11-point numerical rating scale (NRS) for pain, following repeated subcutaneous administration of CAM2038 weekly and CAM2038 monthly in adult opioid-dependent subjects-Safety Population. 11 point scale ranging from 0-10, with 0 being the least amount of pain to 10 being the worst pain imaginable.
Time Frame: 99 days for Group 1, 162 days for Group 2, 127 days for Group 3
Population: Safety Population: included all subjects who received CAM2038. Participants did not always enter pain scores in electronic diaries. Also, participants early terminated during the study and stopped entering scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 32 mg CAM2038 Weekly | 128 mg CAM2038 Monthly Injection | 160 mg CAM2038 Monthly Injection
Number analyzed (Participants) | 28 | 20 | 17
score on a scale
  Baseline: number analyzed (Participants) | 6 | 4 | 16
  Baseline | 7.6 (0.33) | 8.3 (1.30) | 6.1 (2.07)
  Week 1: number analyzed (Participants) | 27 | 19 | 17
  Week 1 | 5.8 (2.40) | 4.9 (2.79) | 5.6 (2.10)
  Week 2: number analyzed (Participants) | 25 | 18 | 15
  Week 2 | 5.4 (2.27) | 5.2 (2.49) | 5.4 (1.85)
  Week 3: number analyzed (Participants) | 24 | 18 | 16
  Week 3 | 5.3 (2.25) | 5.3 (2.77) | 5.4 (2.05)
  Week 4: number analyzed (Participants) | 23 | 18 | 16
  Week 4 | 4.6 (2.23) | 5.5 (2.92) | 5.6 (2.31)
  Week 5: number analyzed (Participants) | 23 | 16 | 15
  Week 5 | 4.8 (2.28) | 4.2 (2.08) | 5.3 (1.88)
  Week 6: number analyzed (Participants) | 22 | 17 | 16
  Week 6 | 4.7 (2.04) | 4.6 (2.70) | 5.2 (1.98)
  Week 7: number analyzed (Participants) | 23 | 17 | 15
  Week 7 | 4.3 (2.11) | 4.9 (2.44) | 5.8 (2.32)
  Week 8: number analyzed (Participants) | 15 | 17 | 14
  Week 8 | 5.2 (1.53) | 5.5 (2.52) | 6.1 (2.08)
  Week 9: number analyzed (Participants) | 14 | 16 | 13
  Week 9 | 5.3 (1.55) | 5.2 (2.73) | 4.9 (2.19)
  Week 10: number analyzed (Participants) | 12 | 15 | 12
  Week 10 | 4.9 (1.69) | 4.8 (2.60) | 5.2 (2.02)
  Week 11: number analyzed (Participants) | 11 | 15 | 11
  Week 11 | 5.2 (1.39) | 4.5 (2.62) | 5.3 (2.32)
  Week 12: number analyzed (Participants) | 10 | 15 | 11
  Week 12 | 5.2 (1.53) | 5.2 (2.30) | 5.9 (2.34)
  Week 13: number analyzed (Participants) | 10 | 15 | 11
  Week 13 | 5.1 (1.58) | 4.4 (2.70) | 4.4 (2.14)
  Week 14: number analyzed (Participants) | 3 | 14 | 10
  Week 14 | 6.4 (3.76) | 4.6 (2.37) | 5.1 (1.96)
  Week 15: number analyzed (Participants) | 0 | 14 | 10
  Week 15 |  | 4.5 (2.54) | 5.5 (2.08)
  Week 16: number analyzed (Participants) | 0 | 12 | 10
  Week 16 |  | 5.5 (2.37) | 5.8 (2.24)
  Week 17: number analyzed (Participants) | 0 | 10 | 3
  Week 17 |  | 5.9 (1.76) | 4.3 (0.76)
  Week 18: number analyzed (Participants) | 0 | 10 | 0
  Week 18 |  | 5.7 (2.13) |
  Week 19: number analyzed (Participants) | 0 | 11 | 0
  Week 19 |  | 5.8 (2.03) |
  Week 20: number analyzed (Participants) | 0 | 9 | 0
  Week 20 |  | 6.3 (1.16) |
  Week 21: number analyzed (Participants) | 0 | 10 | 0
  Week 21 |  | 6.1 (1.61) |
  Week 22: number analyzed (Participants) | 0 | 10 | 0
  Week 22 |  | 5.8 (1.98) |
  Week 23: number analyzed (Participants) | 0 | 1 | 0
  Week 23 |  | 8.0 (NA) — Only one participant entered a pain score, so no SD. |

ADVERSE EVENTS:
Time Frame: 2 years 3 months
Groups:
- 24 mg SL BPN: Group 3: 24 mg Sublingual Buprenorphine (SL BPN) from day 1-7 in group 3
Arm/Group | 32 mg CAM2038 Weekly | 128 mg CAM2038 Monthly Injection | 160 mg CAM2038 Monthly Injection | 24 mg SL BPN
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/20 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/20 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 16/28 | 18/20 | 17/17 | 0/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 32 mg CAM2038 Weekly (N=28) | 128 mg CAM2038 Monthly Injection (N=20) | 160 mg CAM2038 Monthly Injection (N=17) | 24 mg SL BPN (N=18)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Injection Site Swelling (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes Zester (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asparatate aminotransferase inceased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizzyness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tension Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/26/NCT02710526/SAP_000.pdf
  • Study Protocol (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT02710526/Prot_001.pdf